CLINICAL TRIAL: NCT07093671
Title: Mentalization Based Treatment (MBT) in Help Seeking Youths With a Clinical High-Risk Condition for Psychosis (CHR-P): a Randomized Controlled Trial
Brief Title: Mentalization Based Treatment (MBT) in Help Seeking Youths With a Clinical High-Risk Condition for Psychosis (CHR-P)
Acronym: MBT-Psychosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marco Armando (Other)
Responsible Party: Sponsor-Investigator, Marco Armando, PR, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-02579
Record Dates: First submitted 2025-07-07; First posted 2025-07-30 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Psychosis
Keywords: Psychosis; MBT; Mentalization-Based Treatment
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-blinded, superiority, two-arm, parallel group-controlled trial. Participants will be randomized in a 1:1 ratio to either control or intervention group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBCI (No Intervention): Control intervention will consist of routine care based on Need-Based Clinical Intervention (NBCI). All NBCI treatments will be delivered by fully qualified mental health professionals and may include pharmacological treatment, psychotherapeutic sessions, case management, and occupational therapy.
- MBT + NBCI (Experimental): Description: The MBT intervention consists of 24 weekly individual psychotherapy sessions, supplemented by monthly mentalization-based family therapy sessions spread across six phases. The individual sessions are manualized into six blocks, each comprising four weekly sessions. Each block typically begins with sessions that heavily incorporate psychoeducation and progressively transitions to a thematically guided session format. Both patient and family sessions will last 50 minutes, and may be audiotaped for quality control and intern supervision. Participants, along with their families or carers, will be informed of this procedure and retain the right to decline recording. Overall, the program is designed to improve patients' capacity to understand their own and others' mental states and, within interpersonal settings, how these patterns contribute to conflict and psychological distress.
  Interventions: Other: MBT + NBCI

INTERVENTIONS:
Other: MBT + NBCI — The MBT for CHR-P intervention consists of 24 weekly individual psychotherapy sessions, supplemented by monthly mentalization-based family therapy sessions. Both patient and family sessions will last 50 minutes. These psychotherapeutic sessions will complement those received though NBCI by strengthening mentalizing abilities aiming to reduce or prevent detrimental outcomes, by prohibiting or restricting some usual techniques in NBCI treatment (e.g., interpretation, cognitive challenge and Socratic dialogue) and by emphasizing certain techniques (e.g., empathic validation, active management of emotional arousal) which are only sporadically and irregularly used during NBCI treatment. Overall, the program is designed to improve patients' capacity to understand their own and others' mental states and, within interpersonal settings, how these patterns contribute to conflict and psychological distress.
  Arms: MBT + NBCI

SUMMARY:
The primary objective of this study is to evaluate the efficacy of Mentalization-Based Treatment (MBT) combined with Need-Based Clinical Interventions (NBCI) compared to NBCI alone, on CHR-P diagnostic statuses and symptom expression (Hypothesis 1). Specifically, the investigator will assess diagnostic outcomes using a 3-level variable: transition to psychosis, CHR-P status quo, and remission out of CHR-P, as well as CHR-P symptom expression. The investigator hypothesize that: (1a) the experimental treatment (MBT + NBCI) will have a significant effect on diagnostic status (i.e. transition to psychosis) at the end of treatment and follow-up; (1b) the experimental treatment (MBT + NBCI) will significantly reduce the severity of psychotic symptoms at the end of treatment and follow-up.

DETAILED DESCRIPTION:
Schizophrenia incidence peaks between 20 and 24 years, yet approximately one-third of cases manifest before age 18 as Early Onset Psychosis (EOP), which is associated with poorer outcomes compared to adult-onset cases, as reported in most of the literature. Psychoses are among the most severe disorders in children and adolescents (CAD), representing the second leading cause of years lost due to disability worldwide. Evidence suggests that early intervention in psychosis may improve outcomes, and there is increasing consensus among clinicians to initiate treatment as soon as sustained positive psychotic symptoms emerge. Within this early intervention framework, there is a strong hypothesis that intervening during the clinical high risk for psychosis (CHR-P) phase may mitigate, delay, or even prevent the onset of a full psychotic disorder. Reflecting these specific needs, the EPA guidelines recommend psychotherapeutic interventions as the first-line treatment for CHR-P conditions. Despite progress in early identification of psychosis risk states, advancements in psychotherapeutic interventions targeting the so-called "psychosis prodrome" remain limited. Importantly, existing interventions often fall short in addressing predictors of functional outcomes in the long term. Recent psychological, clinical, and neuroscientific studies underscore that socio-emotional difficulties are critical determinants of clinical and functional outcomes in CHR-P individuals. Furthermore, research in social cognition has highlighted that mentalization abilities, which continue to develop through adolescence and into adulthood, depend on complex cerebral connectivity to support functions such as mentalizing, perspective-taking, and moral judgment. These mentalizing processes are fundamental to adult social adaptation and have been shown to play a crucial role in maintaining good mental health. Mentalization-Based Treatment (MBT), a highly effective psychotherapeutic model for addressing socio-emotional difficulties, has been recently adapted for youth at clinical high risk for psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 14-30 years with a CHR-P condition, as defined by the SIPS criteria
* Patients who provide informed consent

Exclusion Criteria:

* Patients with a prior diagnosis of a psychotic disorder
* Intellectual disability (IQ < 70).
* Patients whose psychotic symptoms are primarily induced by substance misuse.
* Patients with significant language barriers
* Parents/legal authority who do not provide informed consent (only minors)
* Adult patient under guardianship

Note: Comorbidities with other psychiatric disorders (e.g., Autism Spectrum Disorder, Personality Disorders) will not constitute an exclusion criterion.

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 212 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
SIPS | At Baseline (T0), at both end of treatment T2 : 24 weeks and at T3 : 48 weeks follow up evaluation
  All primary outcomes will be assessed at baseline (T0) during routine evaluation, end of treatment (T2; 24 weeks), and at 48 weeks follow-up (T3). The primary outcome of this study is the incidence of transition to psychosis within 6 months post-intervention, as measured by the Structured Interview for Psychosis-Risk Syndromes (SIPS). The SIPS is a well-validated, interview-based tool designed to assess symptoms, functioning, and diagnostic criteria for prodromal or at-risk mental states indicative of psychosis. Transition to psychosis, as well as remission from CHR-P state, will be determined based on predefined criteria within the SIPS framework.
  SIPS: Structured Interview for Prodromal Symptoms. Subscales scores (0 to 30). High score = More and/or severe psychotic symptoms

SECONDARY OUTCOMES:
MentS | evaluated at baseline (T0), end of treatment (T2: 24 weeks), and at the T3 (48 weeks follow-up).
  The sub-hypotheses associated with Hypothesis 2 will be assessed using the Mentalization Scale (MentS), which measures three subdomains of mentalizing: self-mentalizing (SM), other-mentalizing (OM), and motivation to mentalize (MM). We will examine both the MentS total score and the three subscale scores independently to test the respective sub-hypotheses.
  MentS: Mentalization Scale. Total score (28 to 140). High score = Better mentalization skills
ETMCQ | evaluated at baseline (T0), end of treatment (T2: 24 weeks), and at the T3 (48 weeks follow-up).
  The sub-hypotheses associated with Hypothesis 3 will be evaluated using the Epistemic Trust, Mistrust, and Credulity Questionnaire (ETMCQ), which includes three subdomains of epistemic trust: trust, mistrust, and credulity. We aim to test the hypotheses using each of the ETMCQ subscale scores separately.
  ETMCQ: Epistemic Trust, Mistrust, and Credulity Questionnaire Subscales scores (5 to 35). "High ""Tust"" score = stronger functional stance of trust High ""Mistrust"" score = stronger maladaptive stances of mistrust High ""Credulity"" score = stronger maladaptive stances of credulity"
GF-R | evaluated at baseline (T0), end of treatment (T2: 24 weeks), and at the T3 (48 weeks follow-up).
  The sub-hypotheses associated with Hypothesis 4 will be examined using the Global Assessment of Functioning - Role (GF-R) scale. These measure is included as part of the SIPS assessment to provide a comprehensive evaluation of role functioning.
  GF-R: Global Functioning - Role scale High score = better functionning
GF-S | evaluated at baseline (T0), end of treatment (T2:24 weeks) and at T3 (48 weeks follow-up)
  The sub-hypotheses associed with Hypothesis 4 will be examined using the Global Assessment of Functioning - Social (GF-S) scale. These measure is included as part of the SIPS assessment to provide a comprehensive evaluation of social functioning.
  GF-S: Global Functioning - Social scale High score = better functionning
MADRS | evaluated at baseline (T0), end of treatment (T2: 24 weeks), and at the T3 (48 weeks follow-up).
  The sub-hypotheses associated with Hypothesis 5 will be assessed using the Montgomery-Asberg Depression Rating Scale (MADRS) 10 items Sum of each item (0 to 60) High score = more severe depressive symptoms
OASIS | evaluated at baseline (T0), end of treatment (T2: 24 weeks), and at the T3 (48 weeks follow-up)
  The sub-hypotheses associated with Hypothesis 5 will be assessed using the Overall Anxiety Severity and Impairment Scale (OASIS).
  5 item, Sum of each item (0 to 20) High score = more severe anxiety symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Marco Armando, PR, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- CHUV, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No